CLINICAL TRIAL: NCT00615199
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center Study To Investigate The Safety And Efficacy Of CP-690,550 In Subjects With Moderate To Severe Crohn's Disease.
Brief Title: A Study to Investigate the Safety and Efficacy of CP-690,550 in Patients With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921043
Record Dates: First submitted 2008-01-14; First posted 2008-02-14 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1mg BD (Experimental)
  Interventions: Drug: CP-690,550
- 5mg BD (Experimental)
  Interventions: Drug: CP-690,550
- 15mg BD (Experimental)
  Interventions: Drug: CP-690,550
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-690,550 — administration via oral route twice daily
  Arms: 1mg BD
Drug: CP-690,550 — administration via oral route twice daily
  Arms: 5mg BD
Drug: CP-690,550 — administration via oral route twice daily
  Arms: 15mg BD
Drug: Placebo — administration via oral route twice daily
  Arms: Placebo BID

SUMMARY:
This study investigates safety and efficacy of CP-690,550 in adult patients with moderate to severe Crohn's disease. The study hypothesis is that at least one of the dose levels to be tested will be more effective than placebo (inactive drug).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age at screening
* Males and females with clinical evidence of Crohn's disease for at least 3 months duration at screening
* Subjects with moderate to severe Crohn's Disease at baseline, as defined by a Crohn's Disease Activity Index (CDAI) score of 220-450 inclusive

Exclusion Criteria:

* Subjects currently receiving immunosuppressants, interferon, anti-TNFa
* Subjects with evidence of hematopoietic disorders
* Subjects with evidence of active or latent TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (64):
- United States (31):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Chevy Chase, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Mexico, Missouri
  - Pfizer Investigational Site, Great Neck, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Upper Saint Clair, Pennsylvania
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Charleston, West Virginia
- Belgium (3):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
- Czechia (2):
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Ústí nad Labem
- France (3):
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy, France
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Pessac
- Hungary (6):
  - Pfizer Investigational Site, Békéscsaba
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Győr
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Kaposvár
  - Pfizer Investigational Site, Szekszárd
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, Amsterdam, Netherlands
- Poland (3):
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Olsztyn
  - Pfizer Investigational Site, Wroclaw
- Slovakia (3):
  - Pfizer Investigational Site, Bratislava, Slovakia
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Nitra
- South Africa (5):
  - Pfizer Investigational Site, Durbanvilee, Cape Town
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Durban, South Africa
  - Pfizer Investigational Site, Cape Town, Western Cape
- Spain (3):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Majadahonda, Madrid
- United Kingdom (2):
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Salford

REFERENCES:
- [Derived] Sandborn WJ, Ghosh S, Panes J, Vranic I, Wang W, Niezychowski W; Study A3921043 Investigators. A phase 2 study of tofacitinib, an oral Janus kinase inhibitor, in patients with Crohn's disease. Clin Gastroenterol Hepatol. 2014 Sep;12(9):1485-93.e2. doi: 10.1016/j.cgh.2014.01.029. Epub 2014 Jan 27. PMID 24480677
- [Derived] Ghoreschi K, Jesson MI, Li X, Lee JL, Ghosh S, Alsup JW, Warner JD, Tanaka M, Steward-Tharp SM, Gadina M, Thomas CJ, Minnerly JC, Storer CE, LaBranche TP, Radi ZA, Dowty ME, Head RD, Meyer DM, Kishore N, O'Shea JJ. Modulation of innate and adaptive immune responses by tofacitinib (CP-690,550). J Immunol. 2011 Apr 1;186(7):4234-43. doi: 10.4049/jimmunol.1003668. Epub 2011 Mar 7. PMID 21383241
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921043&StudyName=A%20Study%20to%20investigate%20the%20safety%20and%20efficacy%20of%20CP-690%2C550%20in%20patients%20with%20moderate%20to%20severe%20Crohn%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet matched to CP-690550 orally twice daily for 4 weeks.
- CP-690550 1 mg: CP-690550 1 milligram (mg) tablet orally twice daily for 4 weeks.
- CP-690550 5 mg: CP-690550 5 mg tablet orally twice daily for 4 weeks.
- CP-690550 15 mg: CP-690550 15 mg tablet orally twice daily for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Started | 34 | 36 | 34 | 35
Completed | 26 | 34 | 33 | 33
Not Completed | 8 | 2 | 1 | 2
Not completed — Adverse Event | 3 | 1 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg | Total
Number analyzed (Participants) | 34 | 36 | 34 | 35 | 139
Age Continuous [Mean (Standard Deviation); unit: years] | 35.7 (12.7) | 36.6 (12.2) | 38.7 (10.2) | 38.1 (11.7) | 37.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 11 | 20 | 17 | 70
  Male | 12 | 25 | 14 | 18 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response 70 at Week 4
Description: Clinical response 70: defined as a reduction in Crohn's Disease Activity Index (CDAI) score from baseline of at least 70 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
Time Frame: Week 4
Population: Full Analysis Set (FAS): all randomized participants who had either withdrawn as treatment failure or completed at least 1 week of dosing and had at least 1 valid CDAI score during the active double-blind phase. Number of participants analyzed excluded those with missing data or who fell outside the visit window.
Measure: Number; unit: participants
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Number analyzed (Participants) | 32 | 35 | 30 | 33
participants | 14 | 13 | 18 | 16

2. Secondary Outcome: Number of Participants With Clinical Response 70 at Week 1 and 2
Description: Clinical response 70: defined as a reduction in CDAI score from baseline of at least 70 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
Time Frame: Week 1, 2
Population: FAS: all randomized participants who had either withdrawn as treatment failure or completed at least (>=)1 week of dosing and had >=1 valid CDAI score during active double-blind phase. Number of participants analyzed excluded those with missing data or who fell outside visit window. 'n'=participants evaluable at given time point for each group.
Measure: Number; unit: participants
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Number analyzed (Participants) | 34 | 36 | 32 | 35
participants
  Week 1 (n=34,36,32,35) | 12 | 9 | 11 | 9
  Week 2 (n=31,36,31,35) | 10 | 15 | 13 | 16

3. Secondary Outcome: Number of Participants Achieving Clinical Remission at Week 4
Description: Clinical remission=CDAI at Week 4 less than (<) 150 points. CDAI is a composite index consisting of a weighted scoring of 8 disease variables:number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI score was based partly on entries (7 days before evaluation) from participant's Diary kept while on study. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
Time Frame: Week 4
Population: FAS: all randomized participants who had either withdrawn as treatment failure or completed at least 1 week of dosing and had at least 1 valid CDAI score during the active double-blind phase. Number of participants analyzed excluded those with missing data or who fell outside the visit window.
Measure: Number; unit: participants
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Number analyzed (Participants) | 32 | 35 | 30 | 33
participants | 7 | 11 | 8 | 5

4. Secondary Outcome: Number of Participants With Clinical Response 100 at Week 4
Description: Clinical response 100: defined as a reduction in CDAI score from baseline of at least 100 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Number analyzed (Participants) | 32 | 35 | 30 | 33
participants | 9 | 11 | 14 | 13

5. Secondary Outcome: Time to First Clinical Remission
Description: Clinical remission=CDAI <150 points. CDAI is a composite index consisting of a weighted scoring of 8 disease variables:number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI score was based partly on entries (7 days before evaluation) from participant's Diary kept while on study. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
Time Frame: Week 1 through Week 4
Population: FAS population: included all randomized participants who had either withdrawn as treatment failure or completed at least 1 week of dosing and had at least 1 valid CDAI score during the active double-blind phase.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Number analyzed (Participants) | 34 | 36 | 33 | 35
days | NA [29.0 to NA] — Median time and upper limit of 95 percent (%) confidence interval (CI) were not estimable as few numbers of participants had remission. | NA [30.0 to NA] — Median time and upper limit of 95% CI were not estimable as few numbers of participants had remission. | 30.0 [30.0 to NA] — Upper limit of 95% CI was not estimable as few numbers of participants had remission. | NA [NA to NA] — Median time and 95% CI were not estimable as few numbers of participants had remission.

6. Secondary Outcome: Time to First Response 70
Description: Clinical response 70: defined as a reduction in CDAI score from baseline of at least 70 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 , higher score indicates higher disease activity.
Time Frame: Week 1 through Week 4
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Number analyzed (Participants) | 34 | 36 | 33 | 35
days | 29.0 [11.0 to 29.0] | 30.0 [15.0 to NA] — Upper limit of 95% CI was not estimable due to insufficient event times. | 21.0 [13.0 to 30.0] | 29.0 [15.0 to NA] — Upper limit of 95% CI was not estimable due to insufficient event times.

7. Secondary Outcome: Time to First Response 100
Description: as for outcome 4
Time Frame: Week 1 through Week 4
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Number analyzed (Participants) | 34 | 36 | 33 | 35
days | NA [28.0 to NA] — Median time and upper limit of 95% CI were not estimable due to insufficient event times. | 30.0 [29.0 to NA] — Upper limit of 95% CI was not estimable due to insufficient event times. | 30.0 [21.0 to NA] — Upper limit of 95% CI was not estimable due to insufficient event times. | NA [16.0 to NA] — Median time and upper limit of 95% CI were not estimable due to insufficient event times.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | CP-690550 1 mg | CP-690550 5 mg | CP-690550 15 mg
Serious Adverse Events (participants affected / at risk) | 5/34 | 4/36 | 4/34 | 1/35
Other Adverse Events (participants affected / at risk) | 20/34 | 18/36 | 19/34 | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | CP-690550 1 mg (N=36) | CP-690550 5 mg (N=34) | CP-690550 15 mg (N=35)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Factitious disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | CP-690550 1 mg (N=36) | CP-690550 5 mg (N=34) | CP-690550 15 mg (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Mucous stools (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 3 | 3
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Plicated tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 3
Asthenia (General disorders) | 3 | 3 | 1 | 1
Chills (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 4 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 3
Tenderness (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood iron decreased (Investigations) | 1 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Faecal calprotectin (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 3 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 3
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0
Anorgasmia (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Factitious disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 2
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 0 | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.